CLINICAL TRIAL: NCT03278730
Title: Phase 2 Single Center, Randomized, Placebo-controlled, Double-blind, Parallel Group Study to Evaluate Efficacy of Para-Tyrosine Supplementation on the Survival and Clinical Outcome in Patients With Sepsis
Brief Title: Efficacy of Para-Tyrosine Supplementation on the Survival and Clinical Outcome in Patients With Sepsis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of resources to start
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, István Wittmann, Professor, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PTE-2015-02
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: sepsis; para-Tyrosine; ortho-Tyrosine; meta-Tyrosine
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: The objective is to evaluate, whether p-Tyr supplementation reduces the ICU mortality of the patients with sepsis comparing to placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Para-Tyrosine intervention (Active Comparator): The patients will receive the study drug during their stay at the ICU but for a maximum of 7 days.
  Study drug will be dispensed by a nominated member of the study team and administered to the patients by the ICU staff via nasogastric tube in form of oral suspension. The content of the hard capsules will be dissolved in 20 ml of tap water before the dosing.
  Drug name: Tyrosine. Strength 500 mg. Oral dose form: hard capsule. Number of Dispensed at frequency of 3x2 g daily. Duration of administration: 4 to 7 days.
  Interventions: Drug: Para-Tyrosine supplementation
- Placebo (Placebo Comparator): The patients will receive the study drug during their stay at the ICU but for a maximum of 7 days.
  Study drug will be dispensed by a nominated member of the study team and administered to the patients by the ICU staff via nasogastric tube in form of oral suspension. The content of the hard capsules will be dissolved in 20 ml of tap water before the dosing.
  Drug name: Placebo.. Strength N/A. Oral dose form: capsule matching to Tyrosine capsule. Number of Dispnsed an frequency 3x2 g daily. Duration of administration: 4 to 7 days.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Para-Tyrosine supplementation — Patients will recieve the study drug during their stay at the ICU, but for a maximum of 7 days. The study drug is 3x2 gramms of para-Tyrosine, which will be dispensed and administered in a form of oral suspension via a nasogastric tube.
  Arms: Para-Tyrosine intervention
Drug: Placebo solution — Patients will recieveplacebo during their stay at the ICU, but for a maximum of 7 days. The study drug is 3x2 gramms of placebo, which will be dispensed and administered in a form of oral suspension via a nasogastric tube.
  Arms: Placebo

SUMMARY:
Meta-and ortho-Tyrosine are known markers of oxidative stress, while the physiological isomer, para-Tyrosine is suggested the antagonize the effects of meta- and ortho-Tyrosine. The changes in the serum levels of meta- and ortho-Tyrosine have been found to be paralel to that of the common sepsis markers. The hypothesis of the study is, that supplementation of para-Tyrosine (p-Tyr) in the early phase of sepsis may diminish some specific inflammatory procedures and thus may have a favourable impact on the disease progress, and consequently on the mortality.

DETAILED DESCRIPTION:
Data suggest, that among the amino acids, the meta- and ortho- isomers of tyrosine are potential markers of oxydative stress. The changes in their serum levels (and urinary excretion) in sepsis were found to be parallel to the changes of the common inflammatory markers, i.e. C-reactive protein (CRP) and pro-calcitonin (PCT). However, para-Tyrosine, which is the isomer physiologically present, seemed to have different kinetics. Furthermore, according to the observations, pathological processes linked to the inflammation could be attenuated or partially or completely reversed by para-tyrosine.

The hypothesis of the study is, that supplementation of para-Tyrosine (p-Tyr) in the early phase of sepsis may diminish some specific inflammatory procedures and thus may have a favourable impact on the disease progress, and consequently on the mortality.

The primary objective of the study is to evaluate, whether oral P-Tyr supplementation reduces mortality compared to placebo group during the ICU stay in patients with sepsis.

The primary endpoint is the comparison of mortality starting from randomization and start of treatment (which should be on the same day) during the period of ICU stay between the active treatment group and placebo group. The secondary objectives of the study are:

to evaluate whether supplementation of p-Tyr has effect on clinical outcome of sepsis compared to placebo in patients receiving appropriate standard care; to evaluate the effect of p-Tyr supplementation on 28-day survival of patients with sepsis; to evaluate, whether the treatment can reduce the time of the ICU stay, to evaluate the effect on overall mortality of patients with sepsis during their hospitalization, to evaluate the effect of p-Tyr supplemetation on the overall hospitalization time, to evaluate the safety of the investigational product. The investigators wish to explore To explore whether serum level of p-Tyr can be maintained with the oral supplementation; dynamics and interrelation of the levels of oxidative stress markers (o- and m-Tyr) and the physiologic isomer of Tyr (p-Tyr) and Phenylalanine (Phe) and the correlation of o-Tyr and m-Tyr serum levels and other parameters of inflammation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria to be eligible for the study:

1. Are able to provide written informed consent (either the patient or the person entitled by legislation to consent on behalf of the patient)
2. Male and female patients ≥ 18 years
3. Have a current primary diagnosis of sepsis based on the the third international consensus definitions for sepsis and septic shock (Sepsis-3)Willing and able to comply with all aspects of the protocol
4. Females of childbearing potential must have negtive serum pregnancy test az screening. (All females will be considered to be of childbearing potential unless they are postmenopausal i.e. amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause or have been sterilized surgically i.e. bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)

Exclusion Criteria:

Subjects must not have any of the following criteria to be eligible for the study:

1. Females who are pregnant (positive β-hCG test at screening) or breastfeeding
2. chronic use of steroids or immunosuppressive drugs within the past 3 months
3. other therapy influencing the immune system within the past 3 months (radiotherapy, chemotherapy etc.)
4. malignant hematologic disease
5. jejunal tube feeding
6. any other significant illness in the medical history ongoing in the preceeding 1 month, which may have an influence on the survival and clinical outcome of the patients (e.g severe chronic heart failure NYHA III-IV., AMI, stroke, major surgery, COPD, renal failure, hepatic failure, hepatic cirrhosis etc.)
7. Life expectancy less, than 1 months according to the judgement of the Investigator (even without significant illness, due to age or general status of the patient)
8. Hypersensitivity to any of the excipients of the study product
9. Known to be human immunodeficiency virus (HIV) positive
10. Active viral hepatitis (B or C) as demonstrated by positive serology
11. History of drug or alcohol dependency or abuse within approximately the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Comparison of mortality starting from randomization and start of treatment (which should be on the same day) during the period of ICU stay between the active treatment group and placebo group.

SECONDARY OUTCOMES:
Effect of para-Tyrosine supplementation on the clinical outcome of sepsis | 30 days
  The investigators wish to evaluate whether supplementation of p-Tyr has effect on clinical outcome (appearance of organ failures due to sepsis: renal failure, respiratory failure, coagulation disorders, hepatic failure, cardiac failure, need for vasopressors, CH balance, nitrogen-balance) of sepsis compared to placebo in patients receiving appropriate standard care. The investigators wish to assess wether para-Tyrosine supplementation can ameliroate the time course and severity of sepsis
Long term effects of para-Tyrosine supplementation on survival | 28 days
  The investigators would like to evaluate the effect of p-Tyr supplementation on 28-day survival of patients with sepsis based on the patients' electronic documentation
Reduction in the time of ICU stay | 30 days
  The investigators shall evaluate, whether the treatment can reduce the time of the ICU stay
Overall mortality | 60 days
  The investigators will evaluate the effect on overall mortality of patients with sepsis during their hospitalization
Hospitalization time | 60 days
  The investigators will evaluate the effect of p-Tyr supplemetation on the overall hospitalization time
Safety and tolerability of para-Tyrosine supplementation (Incidence of Treatment-Emergent Adverse Events) | 60 days
  The investigators wish to evaluate the safety of the investigational product: Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events shall be recorded, using physiological parameters such as impairment in renal and hepatic function, bone marrow toxicity, severe blood pressure changes, tachycardia etc.

OTHER OUTCOMES:
Effect of supplementation on the maintanance of the serum level of para-Tyrosine | 30 days
  The investigators will explore using high performance liquid cromatography (HPLC) whether serum level of p-Tyr can be maintained with the oral supplementation
Assessment of pharmacodynamics | 10 days
  Exploration of the dynamics and interrelation of the levels of oxidative stress markers (o- and m-Tyr) and the physiologic isomer of Tyr (p-Tyr) and Phenylalanine (Phe)
Correlation of o-Tyr and m-Tyr serum levels and other parameters of inflammation | 10 days
  The investigators will assess the correlation of o-Tyr and m-Tyr serum levels and other parameters of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: István Wittmann, MD,PhD,DSc, Principal Investigator — University of Pecs
Locations (2):
- Hungary (2):
  - 2nd Department of Medicine and Nephrological Center, Pécs, Baranya
  - Department of Anaesthesiology and Intensive Care, Pécs, Baranya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brasnyo P, Molnar GA, Mohas M, Marko L, Laczy B, Cseh J, Mikolas E, Szijarto IA, Merei A, Halmai R, Meszaros LG, Sumegi B, Wittmann I. Resveratrol improves insulin sensitivity, reduces oxidative stress and activates the Akt pathway in type 2 diabetic patients. Br J Nutr. 2011 Aug;106(3):383-9. doi: 10.1017/S0007114511000316. Epub 2011 Mar 9. PMID 21385509
- [Background] Bernard GR, Wheeler AP, Russell JA, Schein R, Summer WR, Steinberg KP, Fulkerson WJ, Wright PE, Christman BW, Dupont WD, Higgins SB, Swindell BB. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. N Engl J Med. 1997 Mar 27;336(13):912-8. doi: 10.1056/NEJM199703273361303. PMID 9070471
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Dandona P, Mohanty P, Hamouda W, Ghanim H, Aljada A, Garg R, Kumar V. Inhibitory effect of a two day fast on reactive oxygen species (ROS) generation by leucocytes and plasma ortho-tyrosine and meta-tyrosine concentrations. J Clin Endocrinol Metab. 2001 Jun;86(6):2899-902. doi: 10.1210/jcem.86.6.7745. PMID 11397907
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Druml W, Heinzel G, Kleinberger G. Amino acid kinetics in patients with sepsis. Am J Clin Nutr. 2001 May;73(5):908-13. doi: 10.1093/ajcn/73.5.908. PMID 11333844
- [Background] Hirose T, Shimizu K, Ogura H, Tasaki O, Hamasaki T, Yamano S, Ohnishi M, Kuwagata Y, Shimazu T. Altered balance of the aminogram in patients with sepsis - the relation to mortality. Clin Nutr. 2014 Feb;33(1):179-82. doi: 10.1016/j.clnu.2013.11.017. Epub 2013 Dec 14. PMID 24377412
- [Background] Jensen GL, Miller RH, Talabiska DG, Fish J, Gianferante L. A double-blind, prospective, randomized study of glutamine-enriched compared with standard peptide-based feeding in critically ill patients. Am J Clin Nutr. 1996 Oct;64(4):615-21. doi: 10.1093/ajcn/64.4.615. PMID 8839508
- [Background] Jorres RA, Holz O, Zachgo W, Timm P, Koschyk S, Muller B, Grimminger F, Seeger W, Kelly FJ, Dunster C, Frischer T, Lubec G, Waschewski M, Niendorf A, Magnussen H. The effect of repeated ozone exposures on inflammatory markers in bronchoalveolar lavage fluid and mucosal biopsies. Am J Respir Crit Care Med. 2000 Jun;161(6):1855-61. doi: 10.1164/ajrccm.161.6.9908102. PMID 10852757
- [Background] Kun S, Mikolas E, Molnar GA, Selley E, Laczy B, Csiky B, Kovacs T, Wittmann I. Association of plasma ortho-tyrosine/para-tyrosine ratio with responsiveness of erythropoiesis-stimulating agent in dialyzed patients. Redox Rep. 2014 Sep;19(5):190-8. doi: 10.1179/1351000214Y.0000000090. Epub 2014 Apr 3. PMID 24693974
- [Background] Kun S, Molnar GA, Selley E, Szelig L, Bogar L, Csontos C, Miseta A, Wittmann I. Insulin Therapy of Nondiabetic Septic Patients Is Predicted by para-Tyrosine/Phenylalanine Ratio and by Hydroxyl Radical-Derived Products of Phenylalanine. Oxid Med Cell Longev. 2015;2015:839748. doi: 10.1155/2015/839748. Epub 2015 Oct 20. PMID 26576228
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Liebau F, Sundstrom M, van Loon LJ, Wernerman J, Rooyackers O. Short-term amino acid infusion improves protein balance in critically ill patients. Crit Care. 2015 Mar 12;19(1):106. doi: 10.1186/s13054-015-0844-6. PMID 25882298
- [Background] Lubec B, Hayn M, Denk W, Bauer G. Brain lipid peroxidation and hydroxy radical attack following the intravenous infusion of hydrogen peroxide in an infant. Free Radic Biol Med. 1996;21(2):219-23. doi: 10.1016/0891-5849(96)00018-4. PMID 8818637
- [Background] Mikolas E, Kun S, Laczy B, Molnar GA, Selley E, Koszegi T, Wittmann I. Incorporation of ortho- and meta-tyrosine into cellular proteins leads to erythropoietin-resistance in an erythroid cell line. Kidney Blood Press Res. 2013;38(2-3):217-25. doi: 10.1159/000355770. Epub 2014 Apr 9. PMID 24751667
- [Background] Molnar GA, Nemes V, Biro Z, Ludany A, Wagner Z, Wittmann I. Accumulation of the hydroxyl free radical markers meta-, ortho-tyrosine and DOPA in cataractous lenses is accompanied by a lower protein and phenylalanine content of the water-soluble phase. Free Radic Res. 2005 Dec;39(12):1359-66. doi: 10.1080/10715760500307107. PMID 16298866
- [Background] Molnar GA, Wagner Z, Marko L, Ko Szegi T, Mohas M, Kocsis B, Matus Z, Wagner L, Tamasko M, Mazak I, Laczy B, Nagy J, Wittmann I. Urinary ortho-tyrosine excretion in diabetes mellitus and renal failure: evidence for hydroxyl radical production. Kidney Int. 2005 Nov;68(5):2281-7. doi: 10.1111/j.1523-1755.2005.00687.x. PMID 16221230
- [Background] Szijarto IA, Molnar GA, Mikolas E, Fisi V, Cseh J, Laczy B, Kovacs T, Boddi K, Takatsy A, Gollasch M, Koller A, Wittmann I. Elevated vascular level of ortho-tyrosine contributes to the impairment of insulin-induced arterial relaxation. Horm Metab Res. 2014 Oct;46(11):749-52. doi: 10.1055/s-0034-1387701. Epub 2014 Sep 10. PMID 25208272
- [Background] Molnar GA, Mikolas EZ, Szijarto IA, Kun S, Selley E, Wittmann I. Tyrosine isomers and hormonal signaling: A possible role for the hydroxyl free radical in insulin resistance. World J Diabetes. 2015 Apr 15;6(3):500-7. doi: 10.4239/wjd.v6.i3.500. PMID 25897359
- [Background] Molnar GA, Kun S, Selley E, Kertesz M, Szelig L, Csontos C, Boddi K, Bogar L, Miseta A, Wittmann I. Role of Tyrosine Isomers in Acute and Chronic Diseases Leading to Oxidative Stress - A Review. Curr Med Chem. 2016;23(7):667-85. doi: 10.2174/0929867323666160119094516. PMID 26785996
- [Background] Pandharipande PP, Morandi A, Adams JR, Girard TD, Thompson JL, Shintani AK, Ely EW. Plasma tryptophan and tyrosine levels are independent risk factors for delirium in critically ill patients. Intensive Care Med. 2009 Nov;35(11):1886-92. doi: 10.1007/s00134-009-1573-6. Epub 2009 Jul 9. PMID 19588122
- [Background] Ruggiero RA, Bruzzo J, Chiarella P, di Gianni P, Isturiz MA, Linskens S, Speziale N, Meiss RP, Bustuoabad OD, Pasqualini CD. Tyrosine isomers mediate the classical phenomenon of concomitant tumor resistance. Cancer Res. 2011 Nov 15;71(22):7113-24. doi: 10.1158/0008-5472.CAN-11-0581. PMID 22084446
- [Background] Ruggiero RA, Bruzzo J, Chiarella P, Bustuoabad OD, Meiss RP, Pasqualini CD. Concomitant tumor resistance: the role of tyrosine isomers in the mechanisms of metastases control. Cancer Res. 2012 Mar 1;72(5):1043-50. doi: 10.1158/0008-5472.CAN-11-2964. Epub 2012 Feb 7. PMID 22315349
- [Background] Shaw JH, Wildbore M, Wolfe RR. Whole body protein kinetics in severely septic patients. The response to glucose infusion and total parenteral nutrition. Ann Surg. 1987 Mar;205(3):288-94. doi: 10.1097/00000658-198703000-00012. PMID 3103555
- [Background] Selley E, Kun S, Kurthy M, Kovacs T, Wittmann I, Molnar GA. Para-Tyrosine Supplementation Improves Insulin- and Liraglutide- Induced Vasorelaxation in Cholesterol-Fed Rats. Protein Pept Lett. 2015;22(8):736-42. doi: 10.2174/0929866522666150610093039. PMID 26202368